CLINICAL TRIAL: NCT07247500
Title: Impact of Reventilation After One-Lung Ventilation in Thoracic Surgery (OLVREEXP)
Acronym: OLVREEXP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/0303/HP; 2025-A01698-41 (Other: CHU de Rouen)
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lung Surgery

STUDY DESIGN:
Intervention Model Description: 2 arms in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipulmonary reventilation arm using the accessory circuit (Other): As lobectomy and segmentectomy are procedures of differing complexity, stratification according to the type of surgery will ensure a balanced distribution between the study groups. However, despite their differences, both procedures have similar operative durations and require complete atelectasis of the operated lung. The main distinction lies in the amount of pulmonary parenchyma removed (approximately 10% for segmentectomy and 30% for lobectomy).
  This approach helps minimize bias related to variability in surgical procedures, as lobectomy is generally more invasive than segmentectomy. Consequently, each type of surgery will be represented comparably in both study groups. This stratification ensures that any differences observed between the groups can be attributed to the studied variable rather than to the type of surgical procedure.
  Interventions: Procedure: Bipulmonary Reventilation using the accessory circuit
- Bipulmonary reventilation arm under controlled ventilation (Experimental): As lobectomy and segmentectomy are procedures of differing complexity, stratification according to the type of surgery will ensure a balanced distribution between the study groups. However, despite their differences, both procedures have similar operative durations and require complete atelectasis of the operated lung. The main distinction lies in the amount of pulmonary parenchyma removed (approximately 10% for segmentectomy and 30% for lobectomy).
  This approach helps minimize bias related to variability in surgical procedures, as lobectomy is generally more invasive than segmentectomy. Consequently, each type of surgery will be represented comparably in both study groups. This stratification ensures that any differences observed between the groups can be attributed to the studied variable rather than to the type of surgical procedure.
  Interventions: Procedure: Bipulmonary Reventilation under controlled ventilation

INTERVENTIONS:
Procedure: Bipulmonary Reventilation using the accessory circuit — Bipulmonary Reventilation using the accessory circuit
  Arms: Bipulmonary reventilation arm using the accessory circuit
Procedure: Bipulmonary Reventilation under controlled ventilation — Bipulmonary Reventilation under controlled ventilation
  Arms: Bipulmonary reventilation arm under controlled ventilation

SUMMARY:
Lung cancer is a common disease, and more than 8,000 patients in France undergo lobectomy or pulmonary segmentectomy each year. This surgery remains associated with significant postoperative pulmonary complications, whose incidence ranges from 15% to 49% depending on the study (1). The main complication is pulmonary atelectasis, which provides a favorable setting for the development of postoperative pneumonia.

In thoracic surgery, the operated lung is excluded, and one-lung ventilation is performed on the contralateral lung. During surgery, several strategies exist to prevent atelectasis during one-lung ventilation, known as protective ventilation strategies (2). At the end of the procedure, reventilation allows re-expansion of the previously excluded lung.

However, pulmonary reventilation induces the release of pro-inflammatory cytokines and causes endothelial dysfunction, which may lead to pulmonary edema, thereby negating the benefits of intraoperative protective ventilation. Conversely, insufficient re-expansion may result in persistent postoperative atelectasis, whereas excessive re-expansion can cause volutrauma, alveolar trauma, and/or barotrauma to the operated lung (3).

Several reventilation techniques are currently used, but to our knowledge, the impact of reventilation itself has never been specifically studied. The first, empirical technique, consists of reventilating both lungs using the accessory circuit and the adjustable pressure-limiting (APL) valve, manually bagging the patient over several respiratory cycles (4). The main drawback of this method is the lack of monitoring of insufflated volumes and pressures.

The second, more recent technique, consists of reventilating the patient using the anesthesia machine circuit in controlled ventilation mode, which allows for precise monitoring of pressures and insufflated volumes (5). This approach provides real-time monitoring of lung re-expansion and could therefore be less harmful than the empirical method.

Thus, the objective of this study is to compare postoperative pulmonary complications between patients who underwent lung re-expansion using the accessory circuit and those who underwent lung re-expansion using the anesthesia machine circuit in controlled ventilation mode.

ELIGIBILITY:
Inclusion Criteria:

* ASA score ≤ 3.
* Undergoing a scheduled video-assisted or robot-assisted lobectomy or segmentectomy.
* Patient has read and understood the information sheet and signed the informed consent form.
* For women of childbearing potential, effective contraception and confirmation of the absence of an ongoing pregnancy by a negative blood or urine pregnancy test are required.
* Postmenopausal women (spontaneous, non-medically induced amenorrhea for at least 12 months prior to the inclusion visit).
* Patient affiliated with a social security system.

Exclusion Criteria:

* Patients with a BMI > 40 kg/m².
* Patients with severe chronic respiratory failure (COPD grade 3, FEV₁/FVC < 0.7 and FEV₁ < 50% - according to the GOLD 2025 classification).
* Patients with severe chronic renal failure (GFR < 30 mL/min).
* Patients at high risk of conversion to thoracotomy.
* Patients with a history of acute respiratory distress syndrome (ARDS) within 3 months prior to surgery.
* Patients with a known history of severe hepatic failure (Child-Pugh class B or C).
* Patients with a history of heart failure (NYHA class ≥ II).
* Patients with a history of pulmonary resection.
* Patients with uncontrolled asthma.
* Pregnant or breastfeeding women.
* Patients deprived of liberty by administrative or judicial decision, as well as those under legal protection, guardianship, or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-05-08 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | 7 postoperative days
  The evaluation of the primary endpoint will be performed by an anesthesiologist blinded to the lung re-expansion technique used.
  The composite endpoint will consist of the occurrence, within the first 7 postoperative days, of at least one pulmonary complications (postoperative pneumonia, pleural effusion, postoperative atelectasis, pneumothorax, bronchospasm, or acute respiratory distress syndrome (ARDS)).

SECONDARY OUTCOMES:
Number of postoperative pulmonary complications | 7 postoperative days
  To compare the number of postoperative pulmonary complications between a group of patients who underwent a lung re-expansion technique using the accessory circuit and a group of patients who underwent a lung re-expansion technique using the machine circuit under controlled ventilation.
Number of Death | 30 postopeatives days
  To compare the death level between a group of patients who underwent a lung re-expansion technique using the accessory circuit and a group of patients who underwent a lung re-expansion technique using the machine circuit under controlled ventilation.

IPD SHARING:
Plan to Share IPD: No